CLINICAL TRIAL: NCT06488911
Title: A Phase 3, Open-Label, Long-Term Safety Extension Study Evaluating the Safety and Tolerability of the Fixed-Dose Combination of Obeticholic Acid and Bezafibrate in Subjects With Primary Biliary Cholangitis
Brief Title: To Evaluate Safety and Tolerability of the Fixed- Dose Combination of Obeticholic Acid and Bezafibrate
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Intercept made a business decision to terminate the study based on FDA's request for voluntary withdrawal of Ocaliva and the issuance of clinical hold on studies under US IND involving OCA.
Sponsor: Intercept Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 977-311
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Primary Biliary Cholangitis
Keywords: Primary Biliary Cholangitis; Obeticholic Acid; Bezafibrate; Ursodeoxycholic acid
MeSH Terms: conditions — Liver Cirrhosis, Biliary

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- OCA 5 mg + BZF 400 mg SR (Experimental): Participants will be administered with OCA 5 mg + BZF 400 mg SR once daily.
  Interventions: Drug: FDC tablet (OCA 5 mg + BZF 400 mg SR)

INTERVENTIONS:
Drug: FDC tablet (OCA 5 mg + BZF 400 mg SR) — Participants will be administered with FDC tablets once daily.

SUMMARY:
An Open Label Long-Term Study to Evaluate the Safety and Tolerability of the Fixed-Dose Combination (FDC) of Obeticholic Acid (OCA) and Bezafibrate (BZF) tablet in Subjects with Primary Biliary Cholangitis (PBC).

ELIGIBILITY:
Inclusion Criteria:

* All subjects with PBC who participated and are actively taking investigational product in Study 747-213 or Study 747-214 are eligible to enroll in this study (977-311).

Exclusion Criteria:

* History or presence of other concomitant liver diseases
* Clinical complications of PBC
* History or presence of hepatic decompensating events
* Current or history of gallbladder disease
* If female, known pregnancy, or has a positive urine pregnancy test (confirmed by a positive serum pregnancy test), or lactating.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-10-21 (Actual); Study Completion 2025-10-21 (Actual)

PRIMARY OUTCOMES:
Number of participants reporting adverse events (AE) and serious adverse event (SAE) | Up to 60 months

SECONDARY OUTCOMES:
Number of participants with 50 percent (%) reduction of pruritus determined by visual analogue scale (VAS) score | Up to 60 months
  The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10-centimeter (cm) line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').
Number of participants reporting all-cause mortality | Up to 60 months
Number of participants with Adjudicated Liver Related Clinical Outcomes - Liver transplant | Up to 60 months
Number of participants with Adjudicated Liver Related Clinical Outcomes - Progression to hepatic decompensation | Up to 60 months
Number of participants with Adjudicated Liver Related Clinical Outcomes - Model for End-Stage Liver Disease (MELD) Score ≥15 | Up to 60 months
  MELD is a scoring system for assessing the severity of chronic liver disease and to assess prognosis and suitability for liver transplantation. It uses the participant's values for total bilirubin, serum creatinine, and the international normalized ratio (INR) for prothrombin time to predict survival. MELD score ranges from 6 (less ill) to 40 (gravely ill) with scores and mortality probability being: Score 40=71.3% mortality; Scores 30-39=52.6% mortality; Scores 20-29=19.6% mortality; Scores 10-19=6.0% mortality; Score 9 or less=1.9% mortality. Higher scores indicated greater disease severity. Adjudication was performed under the review of HSAC of all available data for each identified participant to determine liver injury status.

CONTACTS AND LOCATIONS:
Overall Officials: Lynda Szczech, PhD, Study Director — Intercept Pharmaceuticals Inc.
Locations (51):
- United States (13):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Southern California Research Center, Coronado, California
  - Tampa General Medical Group, Tampa, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - NYU Langone Health, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Gastro One, Germantown, Tennessee
  - East Tennessee Research Institute, Johnson City, Tennessee
  - The Liver Institute at Methodist Dallas Medical Center, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - American Research Corporation, San Antonio, Texas
- Argentina (5):
  - DIM Clinica Privada, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - Hospital Italiano de La Plata, Buenos Aires
  - Hospital Universitario Austral, Buenos Aires
  - Hospital Provincial del Centenario, Santa Fe
- Australia (2):
  - Royal Adelaide Hospital, Adelaide
  - Flinders Medical Centre, Bedford Park
- UZ Leuven, Leuven, Belgium
- Canada (2):
  - University of Alberta Division of Gastroenterology Zeidler Ledcor Centre, Edmonton, Alberta
  - Pacific Gastroenterology Associates GI Research Institute, Vancouver, British Columbia
- Universityl Hospital Dubrava, Zagreb, Croatia
- Czechia (3):
  - Hepato-Gastroenterologie HK, s.r.o., Hradec Králové
  - Artroscan s.r.o. Gastroenterologicka, Ostrava
  - Research Site SRO, Pilsen
- Tartu University Hospital, Tartu, Estonia
- France (4):
  - Hopital Henri Mondor, Créteil
  - CHRU de Lille, Lille
  - CHU Paris Est - Hopital Saint Antoine, Paris
  - Hopital de la Pitie Salpetriere, Paris
- Medizinische Hochschule Hannover, Hanover, Germany
- University Hospital of Larissa, Larissa, Greece
- DEOEC II. sz. Belgygyszati Klinika, Debrecen, Hungary
- Hadassah Ein-Karem Medical Center - Liver unit, Jerusalem, Israel
- Azienda Ospedaliero-Universitaria di Bologna Policlinico S. Orsola-Malpighi, Bologna, Italy
- University Hopital Santaros klinikos, Vilnius, Lithuania
- Academisch Medisch Centrum, Amsterdam, Netherlands
- Akershus University Hospital, Lørenskog, Norway
- South Korea (2):
  - Kyungpook National University Hospital, Daegu
  - Seoul National University Bundang Hospital, Seongnam-si
- Spain (2):
  - Hospital ClinicUniversity of Barcelona, Barcelona
  - Consorcio Hospital General Universitario, Valencia
- Turkey (Türkiye) (4):
  - Hacettepe University, Faculty of Medicine, Adult Hospital Gastroenterology, Ankara
  - Ege University, Faculty of Medicine, Gastroenterology, Bornova
  - Istanbul University, Capa Faculty of Medicine, Gastroenterology, Istanbul
  - Harran University Hospital, Gastroenterology, Sanliurfa
- United Kingdom (3):
  - Hull University Teaching Hospitals NHS Trust, Hull
  - Institute of Cellular Medicine Newcastle University, Newcastle upon Tyne
  - John Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No